CLINICAL TRIAL: NCT05824611
Title: Formative Validation of the MoveChecker System
Status: Completed | Type: Observational
Sponsor: Gaia AG (Industry)
Responsible Party: Sponsor
Other Study IDs: MoveChecker Form. Validation
Record Dates: First submitted 2023-03-17; First posted 2023-04-21 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participants: patients with epilepsy included in the study at one of the study locations
  Interventions: Other: collect movement data from epileptic seizures

INTERVENTIONS:
Other: collect movement data from epileptic seizures — non-invasive recording of movement data during care as usual
  Other Names: MoveChecker

SUMMARY:
obtain motion sequences of at least 60 epileptic seizures

DETAILED DESCRIPTION:
Extensive movement data are required to develop an automatic pattern recognition that makes it possible to distinguish movements of epileptic seizures from everyday activities. The aim of collecting formative validation data for the system is to collect movement data from as many epileptic seizures as possible to develop such pattern recognition in the future.

A system is being investigated that uses several non-invasive sensors attached to the extremities and trunk of the test subjects with plasters to record abnormal movement patterns and play them back to detect epileptic seizures with motor involvement. In the study registered here, the movement data of at least 60 epileptic seizures with motor components will be recorded parallel to routine diagnostics using video EEG or video monitoring.

The primary goal is to collect formative validation data for the system. This includes recording the movements of at least 60 epileptic seizures per sample during the hospital stay of the participants to develop future pattern recognition for the system. The secondary goals include the qualitative assessment of the clinical benefit of the system from the point of view of the patient and the medical staff.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* diagnosis of epilepsy (ICD code G40.x)

Exclusion Criteria:

* suspected epilepsy (no diagnosis)
* comorbidities affecting the motor system
* dermatosis in an area of the body relevant to the sensor attachment
* contact allergy due to plaster or sensor material
* known or current illness or disorder that interferes with the ability to understand study participation requirements or to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are included in special care clinics (epilepsy monitoring units), study inclusion is confirmed by a physician at the clinic
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
motion sequences of at least 60 epileptic seizures | up to 4 days
  Motion sequences of at least 60 epileptic seizures, that include the spatial orientation of the nine sensors attached to the participant sampled and recorded at a rate of 30Hz continuously

SECONDARY OUTCOMES:
qualitative assessment of the clinical benefit of the system | through study completion
  Semi-standardised interviews with clinical staff and patients

CONTACTS AND LOCATIONS:
Overall Officials: Michael Domhardt, Dr.-Ing., Principal Investigator — GAIA AG (Sponsor)
Locations (4):
- Germany (4):
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Krankenhaus Mara Universitätsklinikum OWL der Universität Bielefeld, Bielefeld, North Rhine-Westphalia
  - Epilepsiezentrum Kleinwachau, Radeberg, Saxony
  - Evangelisches Krankenhaus Königin Elisabeth Herzberge, Berlin